CLINICAL TRIAL: NCT06439264
Title: Assessing the Clinical Efficacy of Bentonite Clay Gel on Bone Regeneration in the Treatment of Intra-bony Defects: A Clinico-radiograph Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr R Viswa Chandra (Other)
Responsible Party: Sponsor-Investigator, Dr R Viswa Chandra, PROFFESSOR AND HEAD OF THE DEPARTMENT, SVS Institute of Dental Sciences
Organization: SVS Institute of Dental Sciences (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SVSInstituteDS
Record Dates: First submitted 2024-05-17; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Bone Regeneration
MeSH Terms: interventions — Durapatite

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test group (Experimental): In test group, after reflection of flap and degranulation, bone graft i.e., bentonite clay gel with hydroxyapatite will be placed in the void created by the defect and sutures will be placed
  Interventions: Other: bentonite clay gel with hydroxyapatite
- control group (Active Comparator): In control group, after reflection of flap and degranulation, bone graft i.e., hydroxyapatite will be placed in the defect and sutures will be placed.
  Interventions: Other: bentonite clay gel with hydroxyapatite

INTERVENTIONS:
Other: bentonite clay gel with hydroxyapatite — bentonite clay gel presents great potential for bone healing and it leads to the formation of interconnected microporous structure, which can promote native cell infiltration, proliferation,

SUMMARY:
The aim of this study is to evaluate osseous regeneration efficacy of bentonite gel with hydroxyapatite in comparison with hydroxyapatite incase of intrabony defects

The test group includes patients with intrabony defects where flap surgery is will be performed and bentonite clay gel with HA will be placed and in control group only HA is placed.

DETAILED DESCRIPTION:
Experimental: Main treatment group bentonite with hydroxyaatite is added into the defect site.

Comparator: In patients allocated to control group,only hydroxyapatite is added.

ELIGIBILITY:
Inclusion Criteria:

1. Systemically healthy male and female patients of age >18 years
2. two-walled or three-walled intrabony defects and
3. probing pocket depths (PPD) of ≥ 5mm.

Exclusion Criteria:

1. Medically compromised patients,
2. patients <18 years of age,
3. pregnant women,
4. heavy smokers, and
5. patients who underwent radiotherapy or chemotherapy are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
RVG | baseline , 3months,6months
  1. Radiovisiography will be used to assess bone regeneration achieved post operatively after 3 months and 6 months.
probing depth | baseline , 3months,6months
  2. Assessment of probing depth using probe at baseline and postoperatively at 3 and 6 months
clinical attachment level | baseline , 3months,6months
  Assessment of clinical attachment level using probe at baseline and post operatively at 3 and 6 months.

SECONDARY OUTCOMES:
1. Assessment of plaque - according to Turesky modification of Quigley and Hein Plaque Index, 1970. 2. Assessment of Gingivitis - according to Loe H and Silness P, 1963. | baseline ,3months,6months
  1. Assessment of plaque - according to Turesky modification of Quigley and Hein Plaque Index, 1970.
  2. Assessment of Gingivitis - according to Loe H and Silness P, 1963.

CONTACTS AND LOCATIONS:
Locations (1):
- Svs Dental College, Mahbūbnagar, Telangana, India

IPD SHARING:
Plan to Share IPD: No